CLINICAL TRIAL: NCT01701752
Title: A Randomised, Double Blind, Double Observer Study to Assess Repeated Administration of a Single Dose of an Influenza A Vaccine (FP-01.1) Formulated With and Without Adjuvant, in the Presence or Absence of a Single Dose of a Trivalent Inactivated Influenza Virus Vaccine in Subjects 65 to 74 Years of Age.
Brief Title: Influenza A Vaccine (FP-01.1) Formulated With and Without Adjuvant, in the Presence or Absence of a Single Administration of a Trivalent Inactivated Influenza Virus Vaccine in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Targeting Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FP-01.1_CS_03
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Influenza A
Keywords: Influenza A
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Active Comparator): Day 1: FP-01.1 + Placebo ; Day 29: FP-01.1
  Interventions: Biological: FP-01.1 + Placebo; Biological: FP-01.1
- Group 2 (Active Comparator): Day 1: FP-01.1 + TIV ; Day 29: FP-01.1
  Interventions: Biological: FP-01.1 + TIV; Biological: FP-01.1
- Group 3 (Active Comparator): Day 1: FP-01.1-Adjuvant + Placebo ; Day 29: FP-01.1-Adjuvant
  Interventions: Biological: FP-01.1-Adjuvant + Placebo; Biological: FP-01.1-Adjuvant
- Group 4 (Active Comparator): Day 1: FP-01.1-Adjuvant + TIV ; Day 29: FP-01.1-Adjuvant
  Interventions: Biological: FP-01.1-Adjuvant + TIV; Biological: FP-01.1-Adjuvant
- Group 5 (Active Comparator): Day 1: Adjuvant + TIV ; Day 29: Placebo
  Interventions: Biological: Adjuvant + TIV; Other: Placebo
- Group 6 (Active Comparator): Day 1: Placebo + TIV ; Day 29: Placebo
  Interventions: Biological: Placebo + TIV; Other: Placebo

INTERVENTIONS:
Biological: FP-01.1 + Placebo
  Arms: Group 1
Biological: FP-01.1 + TIV
  Arms: Group 2
Biological: FP-01.1-Adjuvant + Placebo
  Arms: Group 3
Biological: FP-01.1-Adjuvant + TIV
  Arms: Group 4
Biological: Adjuvant + TIV
  Arms: Group 5
Biological: Placebo + TIV
  Arms: Group 6
Biological: FP-01.1
  Arms: Group 1; Group 2
Biological: FP-01.1-Adjuvant
  Arms: Group 3; Group 4
Other: Placebo
  Arms: Group 5; Group 6

SUMMARY:
This study will evaluate the safety and immunogenicity of FP-01.1 and FP-01.1 reformulated with an adjuvant (FP-01.1-Adjuvant) in relatively healthy subjects 65 to 74 years of age, subjects that are more representative of the target population. Both formulations will be administered alone or concomitantly with the Trivalent Inactivated Influenza Virus (TIV) vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 to 74 years inclusive at the time of consent
* Female subjects will be post-menopausal (no menses for at least 2 years) and therefore of non-child bearing potential
* Male subjects willing to comply with the applicable contraceptive requirements of the protocol, e.g. must agree to refrain from fathering a child until after the safety follow up visit. Male subjects do not need to use contraception if their partner has been through the menopause, or has had a hysterectomy or bilateral oophorectomy. If a male subject's partner is of child bearing potential, male subjects must agree to use a barrier method (condom) as a method of birth control in addition to any contraceptive measures normally taken by his partner, until after the safety follow up visit.
* Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG and laboratory evaluation (haematology & biochemistry) as assessed by the Investigator in relation to the age of the patient.
* An understanding, ability and willingness to fully comply with study procedures and restrictions
* Ability to provide written, personally signed and dated informed consent to participate in the study.
* The subject has a BMI < 35.

Exclusion Criteria:

* As a result of the medical screening process, the Principal Investigator or Co- Investigator considers the subject unfit for the study.
* Women of child-bearing potential
* Clinically significant , uncontrolled, current, chronic or recurrent disease, as deemed by the Investigator, (e.g. cardiovascular, respiratory, endocrine, renal, liver, gastrointestinal, autoimmune, immune suppression, malignancy or other conditions) that could affect the action, absorption or disposition of the IMP or could affect clinical or laboratory assessments.
* Significant illness as judged by the Principal Investigator or Co-Investigator within 2 weeks of the first dose of IMP.
* Subjects with a history of allergies or allergic conditions including anaphylactic reactions, asthmatics, hay fever, allergy to egg products and eczema sufferers requiring medication which in the opinion of the Principal Investigator or Co- Investigator will affect their participation in the study.
* Subjects receiving medications that affect the immune system including systemic steroids at a dose greater than 5mg and patients on chronic medications where the dose has not been stable for at least 3 months. Inhaled or topical steroids will be allowed.
* Known or suspected intolerance or hypersensitivity to the IMP, or closely related compounds or any of the stated ingredients.
* Male subjects who consume more than 21 units of alcohol per week and female subjects who consume more than 14 units of alcohol per week.
* A positive HIV antibody screen, Hepatitis B surface antigen, Hepatitis B core antibody, or Hepatitis C antibody screen
* Subjects who have significant scarring, tattoos, abrasions, cuts or infections, that in the opinion of the Investigator could interfere with evaluation of injection site local reactions, over the deltoid region of both arms as these will be the dose site.
* Donation of blood or blood products (e.g. plasma, platelets) within 90 days prior to or intention to donate blood during the entire study.
* Use of another investigational medicinal product within 90 days prior to receiving the first dose of IMP or intention to enrol in another clinical study throughout the entire study including the follow up period.
* Subject with suspected recent (≤6 months) experience of influenza-like illness (fever [>37.8ºC] and cough and/or sore throat > 2 days- in the absence of a known cause other than influenza)
* Subjects who have received a flu vaccine in the last 6 months
* Any clinically significant abnormalities, in the opinion of the Principal Investigator or Co-Investigator, on electrocardiograms (ECGs)
* In addition, for each subject, a completed medical history questionnaire will be taken as part of the consented study procedure.

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects reporting solicited local reactions and severity of the local reactions | Day 1- 209
To assess and compare the immunogenicity response between groups | Day 1- 209
  The immunogenicity of two different formulations of FP-01.1 after each vaccine injection in each treated group
Number and proportion of subjects reporting unsolicited AEs and Serious Adverse Events (SAEs) | Day 1- 209
Number and proportion of subjects with abnormal haematology, blood chemistry lab assessments | Day 1- 209
Number and proportion of subjects with abnormal vital signs/ECG assessments | Day 1 - 209

SECONDARY OUTCOMES:
Exploratory immunogenicity tests on samples obtained from subjects | Day 1 -209
To assess the impact of FP-01.1 and FP-01.1-Adjuvant on the immune response to TIV | Day 1-209

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, Professor, Principal Investigator — Centre for Vaccinology, Ghent University Hospital